CLINICAL TRIAL: NCT03670953
Title: A Randomized Controlled Study to Compare the Safety and Efficacy of IPX203 With Immediate-Release Carbidopa-Levodopa in Parkinson's Disease Patients With Motor Fluctuations
Brief Title: A Study to Evaluate the Safety and Efficacy of IPX203 in Parkinson's Disease Participants With Motor Fluctuations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPX203-B16-02; 2018-002233-37 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-09

CONDITIONS: Parkinson's Disease (Disorder)
Keywords: Idiopathic Parkinson's Disease; Lewy Body Parkinson's Disease; Paralysis Agitans; Primary Parkinsonism
MeSH Terms: conditions — Parkinson Disease | interventions — Drugs, Generic; carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double dummy, blinded drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IR CD-LD - Dose Adjustment (Active Comparator): Participants started on the same dose as the pre-study dosing regimen of IR CD-LD and then received dose adjusted IR CD-LD tablets daily orally, for a period of 3 weeks. If the participant was taking controlled release carbidopa-levodopa (CR CD-LD), the CR CD-LD was discontinued and substituted with a 1:1 milligram-equivalent dose of IR CD-LD.
  Interventions: Drug: IR CD-LD
- IPX203 - Dose Conversion (Experimental): Participants received extended release (ER) CD-LD (IPX203) capsules orally, every 6 - 12 hours for a period of 4 weeks at a dose based on their most frequent stable dose of IR CD-LD in dose adjustment period. Participant with most frequent stable dose of 25-100 milligrams (mg) IR CD-LD received 70 - 280 mg IPX203 thrice daily (TID); >25-100 - 37.5-150 mg IR CD-LD received 105-420 mg IPX203 TID; >37.5-150 - 50-200 mg IR CD-LD received 140-560 mg IPX203 TID; >50 - 200 mg IR CD-LD received 175-700 mg IPX203 TID. Participants who received a daily total dose of less than 125-500 mg IR CD-LD in dose adjustment received IPX203 every 12 hours. After initial dose conversion from IR CD-LD to IPX203 as per above mentioned dose conversion schedule, the dose of IPX203 could be further adjusted during the 4 week dose conversion period.
  Interventions: Drug: IPX203 ER CD-LD
- IPX203 - Double-Blind Maintenance (Experimental): Participants received IPX203 capsules orally, every 6 - 12 hours for 13 weeks at a stable dose established at the end of dose conversion period along with placebo matched to IR CD-LD.
  Interventions: Drug: IPX203 ER CD-LD; Other: Placebo Matching IPX203
- IR CD-LD - Double -Blind Maintenance (Active Comparator): Participants received IR CD-LD tablets daily orally, for 13 weeks at a stable dose established at the end of dose adjustment period along with placebo matched to IPX203.
  Interventions: Drug: IR CD-LD; Other: Placebo Matching IR CD-LD

INTERVENTIONS:
Drug: IR CD-LD — Active comparator - IR CD-LD
  Other Names: Generic for Sinemet tablets
  Arms: IR CD-LD - Dose Adjustment; IR CD-LD - Double -Blind Maintenance
Drug: IPX203 ER CD-LD — Investigational formulation - ER CD-LD
  Arms: IPX203 - Dose Conversion; IPX203 - Double-Blind Maintenance
Other: Placebo Matching IPX203 — Double dummy placebo capsules
  Arms: IPX203 - Double-Blind Maintenance
Other: Placebo Matching IR CD-LD — Double dummy placebo tablets
  Arms: IR CD-LD - Double -Blind Maintenance

SUMMARY:
To evaluate the safety and efficacy of IPX203 (carbidopa and levodopa) extended-release capsules (IPX203 ER CD-LD) in comparison to immediate release (IR) CD-LD in the treatment of CD-LD-experienced participants with Parkinson's disease (PD) who have motor fluctuations.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study. The study consisted of a 3-week, open-label IR CD-LD dose adjustment period; a 4-week, open-label period for conversion to IPX203; followed by a 13-week double-blind treatment period with participants randomized in a 1:1 ratio, stratified by center, to receive either IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants diagnosed at age ≥ 40 years with PD, consistent with the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria and who are being treated with stable regimens of CD-LD but experiencing motor fluctuations.
* Able to provide written informed consent prior to the conduct of any study-specific procedures.
* Female participants of childbearing potential must have a negative urine pregnancy test at Screening Visit.
* Negative urine screen for drugs of abuse and negative alcohol breath test at Screening.
* Hoehn and Yahr Stages 1, 2, 3, or 4 in the "On" state (part of Movement Disorders Society version of the Unified Parkinson's Disease Rating Scale [MDS-UPDRS] Part III)
* Agrees to use a medically acceptable method of contraception throughout the study and for 6 weeks after completing the study. Medically acceptable methods of contraception that may be used by the participant and/or partner include but are not limited to: abstinence, oral contraception, NuvaRing or transdermal systems, diaphragm with vaginal spermicide, intrauterine device, condom and partner using vaginal spermicide, surgical sterilization (6 months), progestin implant or injection, or postmenopausal female (no menstrual period for ˃ 2 years) or vasectomy (˃ 6 months).
* Montreal Cognitive Assessment (MoCA) score ≥ 24 at Screening Visit in "On" state.
* Able to differentiate "On" state from "Off" state as determined by at least 75% concordance with a trained rater in "On/Off" ratings for 8 ratings over a 4-hour training period. The concordance must include at least 1 "On" and 1 "Off" rating and must be achieved within two 4-hour training sessions.
* Able and willing to comply with the protocol, including completion of diaries and availability for all study visits.
* Responsive to CD-LD therapy and currently being treated on a stable regimen with CD-LD for at least 4 weeks prior to Visit 1.
* At Screening, the participant has predictable "Off" periods.

Exclusion Criteria:

* Received any investigational medications within 30 days or 5 times the half-life, whichever is longer, prior to Visit 1.
* Female participants who are currently breastfeeding or lactating.
* Had prior neurosurgical treatment for PD or if such procedure is planned or anticipated during the study period.
* Allergic to any excipient in the study drugs.
* History of medical conditions or of a prior surgical procedure that would interfere with LD absorption, such as gastrectomy, proximal small-bowel resection, or bariatric surgery.
* History of upper gastrointestinal hemorrhage in participants with peptic ulcer disease within the past 5 years.
* History of glaucoma with intraocular pressures that are elevated despite appropriate medical management.
* History of seizure or epilepsy and experienced at least 1 seizure during the past 12 months or has not been compliant with medically recommended therapy or visits.
* History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias that are not controlled with medical and/or surgical interventions. A recent (≤ 12 months) history of myocardial infarction with secondary arrhythmias is exclusionary regardless of the therapeutic control.
* History of neuroleptic malignant syndrome or of nontraumatic rhabdomyolysis.
* Liver enzyme values ≥ 2.5 times the upper limit of normal; or history of severe hepatic impairment.
* Serum creatinine level ≥ 1.75 times the upper limit of normal; or requires dialysis at the time of Screening.
* Participant with a history of malignant melanoma or with a suspicious undiagnosed skin lesion which in the opinion of the investigator could be melanoma.
* History of drug or alcohol abuse within the 12 months prior to Screening.
* Received within 4 weeks of Screening or planning to take during participation in the clinical study:
* Any doses of a CR CD-LD apart from a single daily bedtime dose, any doses of Rytary, additional CD (eg, Lodosyn) or benserazide (eg, Serazide), or catechol-O-methyl transferase inhibitors (entacapone or tolcapone) or medications containing these inhibitors (Stalevo),
* Nonselective monoamine oxidase inhibitors (MAOI), apomorphine, or antidopaminergic agents, including antiemetics.
* Employees or family members of the investigator, study site, or sponsor.
* Participants who have previously participated in an IPX203 study.
* Participants who, in the opinion of the clinical investigator, should not participate in the study.
* Based on clinical assessment, participant does not adequately comprehend the terminology needed to complete the PD diary.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Impax Study Director, Study Director — Impax Laboratories, LLC
Locations (108):
- United States (56):
  - Xenoscience, Inc. (102), Phoenix, Arizona
  - St. Joseph's Hospital & Medical Center/ Barrow Neurological Institute (156), Phoenix, Arizona
  - Clinical Trials, Inc. (113), Little Rock, Arkansas
  - University of Arkansas for Medical Sciences (117), Little Rock, Arkansas
  - Loma Linda University Health Care, Department of Neurology (137), Loma Linda, California
  - Keck School of Medicine of USC/University of Southern California (106), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian (134), Newport Beach, California
  - SC3 Research - Pasadena (148), Pasadena, California
  - SC3 Research - Reseda (146), Reseda, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion (120), Aurora, Colorado
  - Rocky Mountain Movement Disorders Center (116), Englewood, Colorado
  - Christiana Care Neurology Specialists (153), Newark, Delaware
  - JEM Research Institute (136), Atlantis, Florida
  - Visionary Investigators Network (168), Aventura, Florida
  - University of Miami-UHealth at Boca Raton (152), Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton (121), Boca Raton, Florida
  - MD Clinical (111), Hallandale, Florida
  - Infinity Clinical Research (104), Hollywood, Florida
  - University of Florida Health Science Center(129), Jacksonville, Florida
  - Neurology Associates, P.A. (125), Maitland, Florida
  - University of Miami (149), Miami, Florida
  - Medical Professional Clinical Research Center, INC (163), Miami, Florida
  - Parkinsons's Disease Treatment Center of Southwest Florida (131), Port Charlotte, Florida
  - Infinity Clinical Research, LLC (105), Sunrise, Florida
  - University of South Florida (114), Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology (174), West Palm Beach, Florida
  - Charter Research (166), Winter Park, Florida
  - Emory Brain Health Center (110), Atlanta, Georgia
  - NeuroStudies.net, LLC (155), Decatur, Georgia
  - Northwestern Medical Group Neurology Clinic(145), Chicago, Illinois
  - Central DuPage Hospital (151), Winfield, Illinois
  - Indiana University Health Neuroscience Center (164), Indianapolis, Indiana
  - University of Kansas Medical Center (118), Kansas City, Kansas
  - Quest Research Institute (103), Farmington Hills, Michigan
  - Henry Ford West Bloomfield Hospital (100), West Bloomfield, Michigan
  - Struthers Parkinson's Center (130), Golden Valley, Minnesota
  - Washington University (109), St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health (142), Las Vegas, Nevada
  - Roseman Medical Research Institute/Roseman Medical Group (154), Las Vegas, Nevada
  - Albany Medical College (139), Albany, New York
  - Mount Sinai West-Department of Neurology(172), New York, New York
  - Wake Forest Baptist Health Sciences (127), Winston-Salem, North Carolina
  - Ucgni (133), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center (123), Cleveland, Ohio
  - Cleveland Clinic (144), Cleveland, Ohio
  - University of Toledo, Gardner-McMaster Parkinson Center (122), Toledo, Ohio
  - Movement Disorder Clinic of Oklahoma (115), Tulsa, Oklahoma
  - Medical University of South Carolina (150), Charleston, South Carolina
  - The Vanderbilt Clinic(158), Nashville, Tennessee
  - Neurology Consultants of Dallas, PA (108), Dallas, Texas
  - University of Texas Southwestern Medical Center (143), Dallas, Texas
  - Houston Methodist Neurological Institute/Movement Disorders Clinic (135), Houston, Texas
  - Inova Medical Group-Neurology I (147), Alexandria, Virginia
  - VCU Health - Neuroscience, Orthopaedic and Wellness Center (124), Henrico, Virginia
  - Booth Gardner Parkinson's Care Center (112), Kirkland, Washington
  - Inland Northwest Research (119), Spokane, Washington
- Czechia (6):
  - Fakultni nemocnice u sv. Anny v Brne, I. neurologicka klinika (704), Brno
  - Neurohk, s.r.o (701), Choceň
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Neurologicka klinika (702), Pardubice
  - Clintrial s.r.o. (703), Prague
  - AXON Clinical, s.r.o. (700), Prague
  - Neurologicka ordinace FORBELI s.r.o.(706), Prague
- France (5):
  - CHU de Clermont-Ferrand - Hopital Gabriel Montpied (404), Clermont-Ferrand
  - CHU de Montpellier, Hopital Gui de Chauliac(405), Montpellier
  - Centre Hospitalier Universitaire de Nice (400), Nice
  - INSERM, Centre d'investigation Clinique 1402, CHU de Poitiers (402), Poitiers
  - Centre d'Investigation Clinique 1436-CHU Purpan-Hopital Pierre Paul Riquet (403), Toulouse
- Germany (8):
  - Curiositas ad sanum, Studien und Beratungs GmbH(311), München, Bavaria
  - Klinikum rechts der lsar der TUM, Klinik und Poliklinik fur Neurologie (303), München, Bavaria
  - Kliniken Beelitz GmbH, Neurologisches Fachkrankenhaus fUr Bewegungsstorungen/Parkinson (300), Beelitz-Heilstätten, Brandenburg
  - Gemeinschaftspraxis Dr. med. Joachim Springub/ Wolfgang Schwarz, Studienzentrum Nord-West (306), Westerstede, Lower Saxony
  - St. Josef-Hospital, Universitatsklinik fur Neurologie, Klinisches Forschungszentrum fur Neurodegeneration (301), Bochum, North Rhine-Westphalia
  - Klinik Haag i. OB, Geriatric Hospital (305), Haag in Oberbayern, Oberbayern (Upper Bavaria)
  - Universitatsklinikum Carl Gustav Carus, Klinik und Poliklinik fur Neurologie (307), Dresden, Saxony
  - Dr. med. REINHARDT Ehret Neurologie Berlin Schlobstr. 29 (309), Berlin
- Italy (8):
  - Department "G.F. Ingrassia" Section of neuroscience-Policlinico "Vittorio Emanuele" (608), Catania, Italy/Catania/Sicily
  - Universita G. D'annunzio CeSi Met (604), Chieti, Italy/Chieti/Abbruzzo
  - Centro Ricerca Parkinson San Raffaele Cassino (601), Cassino, Italy/Frosinone/Lazio
  - Fondazione lstituto Neurologico Nazionale "C. Mondino" (606), Pavia, Italy/Pavia/Lombardia
  - Azienda Ospedaliero-Universitaria Pisana (602), Pisa, Italy/Pisa/Toscana
  - University of Rome Tor Vergata/Hospital Tor Vergata (605), Roma, Italy/Roma/Lazio
  - IRCCS San Raffaele Pisana (600), Roma, Italy/Roma/Lazio
  - Department of Neuroscience, Mental Health and Sensory System (NeSMOS), Sapienza University (603), Roma, Italy/Roma/Lazio
- Poland (7):
  - Centrum Medyczne Neuromed (803), Bydgoszcz
  - Szpital Sw. Rozy (805), Krakow
  - Krakowska Akademia Neurologii Sp. z o.o.(802), Krakow
  - NZOZ Neuromed M. i M Nastaj Spolka Partnerska(800), Lublin
  - NZOZ Neuro-Kard Ilkowski i Partnerzy Spolka Partnerska Lekarzy (801), Poznan
  - Neuro-Care Sp. z o.o. sp. k.(804), Siemianowice Śląskie
  - Centrum Medyczne NeuroProtect (806), Warsaw
- Spain (15):
  - Hospital Genral Universitario de Elche (509), Elche, Alicante
  - Hospital Universitari General de Catalunya (504), Sant Cugat del Vallès, Barcelona
  - Hospital Universitari Mutua Terrassa (506), Terrassa, Barcelona
  - Policlinica Gipuzkoa, S.A.,(511), Donostia / San Sebastian, Gipuzkoa
  - Clinica Universidad de Navarra (512), Pamplona, Navarre
  - Hospital Universitario Quiron Dexeus (501), Barcelona
  - Hospital Universitario Vall d' Hebron (505), Barcelona
  - Hospitalaries Del Sagrat Cor De Jesus Hospital Sant Rafael (516), Barcelona
  - Hospital Clinic de Barcelona (507), Barcelona
  - Hospital De La Santa Creu i Sant Pau (502), Barcelona
  - Hospital Universitario de la Princesa (508), Madrid
  - Hospital Universitario Ramon y Cajal (500), Madrid
  - Hospital Universitario Infanta Sofia (513), Madrid
  - Hospital Universitario Virgen del Rocio (503), Seville
  - Hospital Universitario y politecnico La Fe (515), Valencia
- United Kingdom (3):
  - Re: Cognition Health Ltd(205), Plymouth, Devon
  - Re:Cognition Health Ltd (202), London
  - Imperial College Healthcare NHS Trust (200), London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauser RA, Espay AJ, Ellenbogen AL, Fernandez HH, Isaacson SH, LeWitt PA, Ondo WG, Pahwa R, Schwarz J, Stocchi F, Zeitlin L, Banisadr G, Fisher S, Visser H, D'Souza R. IPX203 vs Immediate-Release Carbidopa-Levodopa for the Treatment of Motor Fluctuations in Parkinson Disease: The RISE-PD Randomized Clinical Trial. JAMA Neurol. 2023 Oct 1;80(10):1062-1069. doi: 10.1001/jamaneurol.2023.2679. PMID 37578800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 630 enrolled participants entered the immediate release carbidopa-levodopa (IR CD-LD) dose adjustment period of which 589 participants entered IPX203 conversion period of which 506 participants entered double-blind maintenance period. Participants were randomized in a 1:1 ratio in double blind period.
Pre-assignment Details: Participants with parkinsons disease (PD) who were treated with stable regimens of carbidopa - levodopa (CD - LD) were enrolled in this study.
Period: Dose Adjustment (Weeks 1- 3)
Arm/Group | IR CD-LD - Dose Adjustment | IPX203 - Dose Conversion | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Started | 630 | 0 | 0 | 0
Completed | 589 | 0 | 0 | 0
Not Completed | 41 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0
Not completed — Miscellaneous | 21 | 0 | 0 | 0
Period: Dose Conversion (Weeks 4 - 7)
Arm/Group | IR CD-LD - Dose Adjustment | IPX203 - Dose Conversion | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Started | 0 (Participants who completed dose adjustment period entered the dose conversion period.) | 589 (Participants who completed dose adjustment period started the dose conversion period.) | 0 | 0
Completed | 0 | 506 | 0 | 0
Not Completed | 0 | 83 | 0 | 0
Not completed — Adverse Event | 0 | 35 | 0 | 0
Not completed — Lack of Efficacy | 0 | 10 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Non compliance | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 32 | 0 | 0
Not completed — Miscellaneous | 0 | 2 | 0 | 0
Period: Double Blind Maintenance (Weeks 8 - 20)
Arm/Group | IR CD-LD - Dose Adjustment | IPX203 - Dose Conversion | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Started | 0 | 0 (Participants who completed the dose conversion period were randomized to start double blind period) | 256 (Participants who completed the dose conversion period were randomized to start double blind period) | 250 (Participants who completed the dose conversion period were randomized to start double blind period)
Completed | 0 | 0 | 222 | 227
Not Completed | 0 | 0 | 34 | 23
Not completed — Adverse Event | 0 | 0 | 14 | 3
Not completed — Lack of Efficacy | 0 | 0 | 5 | 8
Not completed — Protocol Violation | 0 | 0 | 3 | 1
Not completed — Non compliance | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 10 | 11
Not completed — Miscellaneous | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were treated with any study drug.
Groups:
- IR CD-LD - Double -Blind Maintenance: Participants received IR CD - LD tablets daily orally, for 13 weeks at a stable dose established at the end of dose adjustment period along with placebo matched to IPX203.
- Not Randomized: Participants who discontinued from dose adjustment and dose conversion.
- Total: Total of all reporting groups
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance | Not Randomized | Total
Number analyzed (Participants) | 256 | 250 | 124 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.02) | 66.5 (8.85) | 67.3 (9.00) | 66.5 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 73 | 64 | 234
  Male | 159 | 177 | 60 | 396
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 31 | 14 | 77
  Not Hispanic or Latino | 223 | 215 | 106 | 544
  Unknown or Not Reported | 1 | 4 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 5 | 3 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 6
  White | 244 | 242 | 120 | 606
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in "Good on" Time Per Day at Week 20/Early Termination (ET)
Description: "Good on" time was derived from the 3-day PD Diaries. For each day, "Good on" time was calculated by adding the number of half-hour intervals in which either an "On" without dyskinesia or "On" with nontroublesome dyskinesia was checked.
  Baseline was defined as data obtained from PD Diary collected over 3 days prior to Week 7/Randomization.
  Least square mean (LSM), standard error (SE), confidence interval (CI), Mixed model repeated measures (MMRM), Change from baseline (CFB).
Time Frame: Baseline (Week 7) and Week 20/ET
Population: The Modified Intent-to-Treat (mITT) Analysis Set included all participants who were randomized and treated and had a valid baseline PD Diary and at least one valid post-randomization PD Diary. Participants with available data at specified time point were included in analysis. Data was planned to be reported only for double-blind Maintenance period.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Number analyzed (Participants) | 249 | 246
hours/day
  Baseline (Week 7) | 11.67 (2.943) | 11.72 (2.759)
  Change at Week 20/ET: number analyzed (Participants) | 235 | 241
  Change at Week 20/ET | -0.39 (2.706) | -0.97 (3.081)
Statistical Analysis 1: Comparison: IPX203 - Double-Blind Maintenance vs IR CD-LD - Double -Blind Maintenance; Test type: Superiority — 2-sided at a significance level of alpha = 0.05; p = 0.0194, MMRM — LSM, SE, CI and p-value from a MMRM with CFB in "Good on" time as outcome, baseline "Good on" time as a covariate, treatment and visit as fixed effects, pooled center as random effect and a treatment-by-visit interaction; The degree-of-freedom of the denominator is estimated using the Kenward-Roger method. Unstructured covariance structure is assumed; Least Squares Mean difference = 0.53, 95% CI 2-sided [0.09 to 0.97], Standard Error of Mean 0.226

2. Secondary Outcome: Change From Baseline in "Off" Time Per Day at Week 20/ET
Description: "Off" time was derived from the 3-day PD Diaries. For each day, "Off" time was calculated by adding the number of half-hour intervals in which the Status "Off" was checked. Baseline was defined as data obtained from PD Diary collected over 3 days prior to Week 7/Randomization.
Time Frame: Baseline (Week 7) and Week 20/ET
Population: mITT population with available data at specified time point. Data was planned to be reported only for double-blind Maintenance period.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Number analyzed (Participants) | 249 | 246
hours/day
  Baseline (Week 7) | 3.95 (2.524) | 4.02 (2.466)
  Change at Week 20/ET: number analyzed (Participants) | 235 | 241
  Change at Week 20/ET | 0.29 (2.235) | 0.76 (2.901)
Statistical Analysis 1: Comparison: IPX203 - Double-Blind Maintenance vs IR CD-LD - Double -Blind Maintenance; Test type: Superiority — 2-sided at a significance level of alpha = 0.05; p = 0.0252, MMRM — LSM, SE, CI and p-value from a MMRM with CFB in "Off" time as outcome, baseline "Off" time as a covariate, treatment and visit as fixed effects, pooled center as random effect and a treatment-by-visit interaction; [statistical method as in outcome 1, analysis 1]; Least Squares Mean difference = -0.48, 95% CI 2-sided [-0.90 to -0.06], Standard Error of Mean 0.214

3. Secondary Outcome: Percentage of Participants With Either "Much Improved" or "Very Much Improved" in Patient Global Impression of Change (PGI-C) Scores at Week 20/ET
Description: The Patient Global Impression of Change (PGIC) is self assessment questionnaire which was used by participants to compare his/her condition on a 7-point scale ranging from 1-Very Much Worse, 2-Much Worse, 3-Minimally Worse, 4-No Change, 5-Minimally Improved, 6-Much Improved, 7-Very Much Improved. Percentage of participants with either "Much Improved" or "Very Much Improved" was reported.
Time Frame: Week 20/ET
Population: The Intent-to-treat (ITT) Analysis Set included all participants who were randomized and treated with any study drug and had a baseline and at least one post-baseline efficacy assessment.
Measure: Number; unit: percentage of participants
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Number analyzed (Participants) | 256 | 250
percentage of participants | 29.7 | 18.8
Statistical Analysis 1: Comparison: IPX203 - Double-Blind Maintenance vs IR CD-LD - Double -Blind Maintenance; Test type: Superiority — 2-sided at a significance level of alpha = 0.05; p = 0.0015, Cochran-Mantel-Haenszel — P-value from the Cochran-Mantel-Haenszel test stratified by pooled center comparing the percentage of "Much" or "Very Much Improved" participants between the treatment groups; Percent difference = 10.9, 95% CI 2-sided [3.5 to 18.3]

4. Secondary Outcome: Change From Baseline in The Movement Disorders Society Version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III at Week 20/ET
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 34 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-234). Part III score ranges from 0 to 136. A higher score indicated more severe symptoms of PD. Baseline was defined as data obtained from PD Diary collected over 3 days prior to Week 7/Randomization.
Time Frame: Baseline (Week 7) and Week 20/ET
Population: ITT population with available data at specified time point. Data was planned to be reported only for double-blind Maintenance period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- IPX203 - Double-Blind Maintenance: Participants received IPX203 capsules orally, every 6 -12 hours for 13 weeks at a stable dose established at the end of dose conversion period along with placebo matched to IR CD-LD.
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Number analyzed (Participants) | 256 | 250
score on a scale
  Baseline (Week 7) | 26.9 (16.62) | 27.0 (16.83)
  Change at Week 20/ET: number analyzed (Participants) | 254 | 249
  Change at Week 20/ET | 1.1 (11.07) | 0.9 (10.10)
Statistical Analysis 1: Comparison: IPX203 - Double-Blind Maintenance vs IR CD-LD - Double -Blind Maintenance; Test type: Superiority — 2-sided at a significance level of alpha = 0.05; p = 0.9587, MMRM — LSM, SE, CI and p-value from a MMRM with CFB in MDS-UPDRS Part III Score as outcome, baseline MDS-UPDRS Part III Score as a covariate, treatment and visit as fixed effects, pooled center as random effect and a treatment-by-visit interaction; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-1.8 to 1.7], Standard Error of Mean 0.89

5. Secondary Outcome: Change From Baseline in The Sum of MDS-UPDRS Part II and Part III at Week 20/ET
Description: MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. (Part I; 13 items) non-motor experiences of daily living, (Part II; 13 items) motor experiences of daily living completed by the participants, (Part III; 34 items) motor examination of PD and was administered by the rater, and (Part IV; 6 items) motor complication integrates participant-derived information with the rater's clinical observations and judgements and is completed by the rater. For each question a numeric score was assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Total Score equals the sum of Parts I, II, and III and IV (Range 0-234). The scale range for Part II+III score is 0-188. A higher score indicated more severe symptoms of PD. Baseline was defined as data obtained from PD Diary collected over 3 days prior to Week 7/Randomization.
Time Frame: Baseline (Week 7) and Week 20/ET
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
Number analyzed (Participants) | 256 | 250
score on a scale
  Baseline (Week 7) | 38.9 (22.20) | 39.3 (21.65)
  Change at Week 20/ET: number analyzed (Participants) | 253 | 248
  Change at Week 20/ET | 2.0 (13.54) | 1.8 (12.39)
Statistical Analysis 1: Comparison: IPX203 - Double-Blind Maintenance vs IR CD-LD - Double -Blind Maintenance; Test type: Superiority — 2-sided at a significance level of alpha = 0.05; p = 0.9668, MMRM — LSM, SE, CI & p-value from MMRM with CFB in MDS-UPDRS Part II & III Scores as outcome, baseline MDS-UPDRS Part II and III Scores as a covariate, treatment and visit as fixed effects, pooled center as random effect & a treatment-by-visit interaction; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.0, 95% CI 2-sided [-2.2 to 2.1], Standard Error of Mean 1.11

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose (Up to Weeks 24)
Groups:
- IR CD-LD - Dose Adjustment: Participants started on the same dose as the pre-study dosing regimen of IR CD-LD and then received dose adjusted IR CD-LD tablets daily orally, for a period of 3 weeks. If the participant was taking CR CD-LD, the CR CD-LD was discontinued and substituted with a 1:1 milligram-equivalent dose of IR CD-LD.
- IPX203 - Dose Conversion: Participants received IPX203 capsules orally, every 6 - 12 hours for a period of 4 weeks at a dose based on their most frequent stable dose of IR CD-LD in dose adjustment period. Participant with most frequent stable dose of 25-100 mg IR CD-LD received 70 - 280 mg IPX203 TID; >25-100 - 37.5-150 mg IR CD-LD received 105-420 mg IPX203 TID; >37.5-150 - 50-200 mg IR CD-LD received 140-560 mg IPX203 TID; >50 - 200 mg IR CD-LD received 175-700 mg IPX203 TID. Participants who received a daily total dose of less than 125-500 mg IR CD-LD in dose adjustment received IPX203 every 12 hours. After initial dose conversion from IR CD-LD to IPX203 as per above mentioned dose conversion schedule, the dose of IPX203 could be further adjusted during the 4 week dose conversion period.
Arm/Group | IR CD-LD - Dose Adjustment | IPX203 - Dose Conversion | IPX203 - Double-Blind Maintenance | IR CD-LD - Double -Blind Maintenance
All-Cause Mortality (participants affected / at risk) | 0/630 | 0/589 | 0/256 | 0/250
Serious Adverse Events (participants affected / at risk) | 7/630 | 12/589 | 8/256 | 4/250
Other Adverse Events (participants affected / at risk) | 40/630 | 130/589 | 35/256 | 32/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IR CD-LD - Dose Adjustment (N=630) | IPX203 - Dose Conversion (N=589) | IPX203 - Double-Blind Maintenance (N=256) | IR CD-LD - Double -Blind Maintenance (N=250)
Anameia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radiation neuropathy (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ejection fraction descreased (Investigations) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
On and off phenomenon (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0
Vertebral artery aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IR CD-LD - Dose Adjustment (N=630) | IPX203 - Dose Conversion (N=589) | IPX203 - Double-Blind Maintenance (N=256) | IR CD-LD - Double -Blind Maintenance (N=250)
Constipation (Gastrointestinal disorders) | 7 | 12 | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 25 | 3 | 2
Nausea (Gastrointestinal disorders) | 7 | 29 | 11 | 2
Vomiting (Gastrointestinal disorders) | 3 | 13 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 13 | 5 | 9
Dizziness (Nervous system disorders) | 3 | 17 | 6 | 2
Dyskinesia (Nervous system disorders) | 11 | 40 | 5 | 1
Insomnia (Psychiatric disorders) | 6 | 13 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 7 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2 | 7
Anxiety (Psychiatric disorders) | 1 | 9 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03670953/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT03670953/SAP_001.pdf